CLINICAL TRIAL: NCT03914534
Title: Bioequivalence Study of Sodium Divalproate Tablets 500 mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tecnoquimicas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Versión 1- BIO 088
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Formulation of Valproic Acid (Experimental): Valproic Acid tablets 500 mg Single dose administered in dosing period 1 or 2
  Interventions: Drug: Valproic Acid 500 MG
- Reference Formulation of Valproic Acid (Active Comparator): Valcote tablets 500 mg Single dose administered in dosing period 1 or 2
  Interventions: Drug: Valcote 500 mg

INTERVENTIONS:
Drug: Valproic Acid 500 MG — Administration of 500 mg of Valproic Acid
  Arms: Test Formulation of Valproic Acid
Drug: Valcote 500 mg — Administration of 500 mg of Valproic Acid
  Arms: Reference Formulation of Valproic Acid

SUMMARY:
The objective of this study is to establish the bioequivalence of two valproic acid formulations through the estimation of valproic acid in plasma samples, according to Food and Drugs Administration (FDA), World Health Organization (WHO) and Colombian National Vigilance Institute for Drugs and Food (INVIMA) guidelines.

DETAILED DESCRIPTION:
This will be a single-center, open-label, four-period, two-treatment, two-sequence, randomized, single-dose, crossover study. 30 healthy adults will be randomized to receive a single dose (500 mg) of the test formulation of valproic acid and reference formulation of valproic acid separately in each treatment period. There will be two treatment sequences (AB, BA) and a 7 day washout between the two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women from 18 to 50 years old
* Diagnosed as healthy after a clinical examination
* BMI from 18 to 30 kg/m2
* Not smoking for at least 3 months
* To sign the informed consent
* Not having participated in a similar study for at least 4 months

Exclusion Criteria:

* Renal, cardiac immunological, dermatological, endocrine, gastrointestinal, neurological or psychiatric condition
* Hematologic disorders, specially anemia and polycythemia
* Permanent or temporal pharmacological therapy, prescribed or not
* Smoking for the last 3 months
* Alcohol drinker more than once a week
* Drug abuse
* Drug hypersensitivity
* Angioedema or anaphylaxis history
* Pregnancy or breast-feeding
* HIV o Hepatitis B diagnosed
* Blood donor in the past 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
(AUC) Area Under the Curve 0-48 | From 0 to 48 hours
  0, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 y 48 hours
Cmax | From 0 to 48 hours
  0, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 y 48 hours

SECONDARY OUTCOMES:
Tmax | From 0 to 48 hours
  0, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 y 48 hours
Kel | From 0 to 48 hours
  0, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 y 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de la Sabana, Chía, Colombia